CLINICAL TRIAL: NCT02250586
Title: Internet Based Cognitive-behavioral Therapy for Concerned Significant Others of Problem Gamblers: a Randomized Wait-list Controlled Trial
Brief Title: Internet Based Cognitive Behavior Therapy for Concerned Significant Others of Problem Gamblers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stockholm University (Other)
Collaborators: Karolinska Institutet (Other); Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Per Carlbring, Professor, Stockholm University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBT-CSO-Gambling
Record Dates: First submitted 2014-09-18; First posted 2014-09-26 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Gambling
Keywords: concerned significant other; internet-delivered cognitive-behavioral therapy,; treatment-refusing problem gambler
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT-CSO (Experimental): The CBT-CSO program will be based on concepts from cognitive-behavioral therapy and motivational interviewing, and is specifically developed for use with CSOs of treatment refusing problem gamblers. The program resembles the community reinforcement and family training approach that has been successfully used with CSOs of substance abusers.
  The program will be given as guided self-help with guidance given via email and telephone. There are 8 modules, which all contain homework exercises and about 5-10 pages of text.
  Interventions: Behavioral: CBT-CSO
- Wait-list (No Intervention): The participants allocated to the control condition will be put on a waiting list and offered the CBT-CSO program after 10 weeks. The CSOs will receive information about available treatment options-in their area and web-based-for the problem gambler.

INTERVENTIONS:
Behavioral: CBT-CSO — Internet-delivered cognitive-behavioral therapy for CSO's of treatment refusing problem gamblers
  Arms: CBT-CSO

SUMMARY:
BACKGROUND: About 2.3 % of the adult population in Sweden is considered to be problem gamblers, and it is estimated that only 5 % of them seek treatment. Problem gambling can have devastating effects on the economy, health and relationship, both for the problem gambler and their concerned significant other (CSO). No empirically supported program exists for the CSOs of problem gamblers. Consequently, the aim of this study is to develop and evaluate a program aimed at CSOs of treatment refusing problem gamblers. The program will be based on principles from cognitive behavioral therapy and motivational interviewing. In order to benefit as many CSOs as possible, the program will be delivered via the Internet with therapist support via email and telephone.

METHODS/DESIGN: This will be a randomized wait-list controlled internet-delivered trial. A cognitive behavioral-therapy program for the concerned significant others (CSOs) of problem gamblers (PGs) will be developed and evaluated. The participants will work through 8 modules over 10 weeks in a secure online environment, and receive support via text messages and over telephone. 150 CSOs over 18 years of age will be included. Measures will be taken at baseline 3, 6 and 12 months. Primary outcomes concern gambling-related harm and motivating the PG to seek treatment. Secondary outcomes are CSO's feelings of depression, anxiety, relationship satisfaction and quality of life.

HYPOTHESIS: The investigators hypothesize: 1) that the CBT-CSO group will lead to a reduction in gambling related harm experienced by the CSO, 2) the CBT-CSO program will reduce the CSO's anxiety and depressive feelings, 3) the CBT-CSO program will decrease the amount of time and money the problem gambler spend on gambling, 4) the CBT-CSO program will increase the CSO's relationship satisfaction with the problem gambler.

ELIGIBILITY:
Inclusion Criteria:

* The CSO and the gambler are at least 18 years old,
* The CSO is a parent, child, sibling, friend or partner of the gambler.
* The CSO must have had a relationship with the gambler for at least 3 months.
* Neither the CSO nor the gambler has had any treatment in the past 3 months (that is related to gambling).
* The gambler is currently refusing help.
* The CSO is able to read and answer questions in Swedish, and is willing to talk to a counselor each week.
* The gambler is a problem gambler according to Problem Gambling Severity Index, as rated by the CSO.
* The CSO must agree to have their telephone calls recorded.

Exclusion Criteria:

* Presence of psychotic- or bipolar disorder in the CSO or gambler.
* CSO meets PGSI criteria for ongoing problem gambling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Inventory of Consequences Scale for the Gambler and CSO | Change from baseline at: [1] end of treatment period; follow-ups at [2] month 6 and [3] month 12 after the treatment period.

SECONDARY OUTCOMES:
9-item Patient Health Questionnaire (PHQ-9) | Change from baseline at: [1] end of treatment period; follow-ups at [2] month 6 and [3] month 12 after the treatment period.
The Generalised Anxiety Disorder 7-item (GAD-7) | Change from baseline at: [1] end of treatment period; follow-ups at [2] month 6 and [3] month 12 after the treatment period.
Relationship Assessment Scale (generic version) | Change from baseline at: [1] end of treatment period; follow-ups at [2] month 6 and [3] month 12 after the treatment period.
WHO Quality of Life Questionnaire-Bref | Change from baseline at: [1] end of treatment period; follow-ups at [2] month 6 and [3] month 12 after the treatment period.
Timeline followback method | Change from baseline at: [1] end of treatment period; follow-ups at [2] month 6 and [3] month 12 after the treatment period.
  CSOs will be asked to report the amount of money spent on gambling by the identified problem gambler.
Treatment engagement | Change from baseline at: [1] end of treatment period; follow-ups at [2] month 6 and [3] month 12 after the treatment period.
  CSO will be asked to report if and when the identified problem gambler enter treatment. "Entering treatment" is defined as attending at least 1 session or calling the National Gambling Helpline

CONTACTS AND LOCATIONS:
Locations (1):
- Stockholm University, Stockholm, Sweden

REFERENCES:
- [Background] Magnusson K, Nilsson A, Hellner Gumpert C, Andersson G, Carlbring P. Internet-delivered cognitive-behavioural therapy for concerned significant others of people with problem gambling: study protocol for a randomised wait-list controlled trial. BMJ Open. 2015 Dec 9;5(12):e008724. doi: 10.1136/bmjopen-2015-008724. PMID 26656017
- [Result] Magnusson K, Nilsson A, Andersson G, Hellner C, Carlbring P. Internet-delivered cognitive-behavioral therapy for significant others of treatment-refusing problem gamblers: A randomized wait-list controlled trial. J Consult Clin Psychol. 2019 Sep;87(9):802-814. doi: 10.1037/ccp0000425. PMID 31403816
- See also: Public website to convey study information and recruitment — https://spel.iterapi.se
- Available data/document: Individual Participant Data Set: awtg7 — https://osf.io — The trial's outcome data and scripts are available for download: https://osf.io/awtg7/